CLINICAL TRIAL: NCT06307405
Title: To Explore the Application of mNGS Detection Technology in the Diagnosis of Pulmonary Infection
Brief Title: The Value of mNGS in Diagnosis of Pulmonary Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Yunfeng Hou (Other)
Responsible Party: Sponsor-Investigator, Yunfeng Hou, associate chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: WJP2023
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Infection
Keywords: Metagenomic next-generation sequencing，Pulmonary Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pulmonry infection group: 50 cases of suspected pulmonary infection (based on clinical manifestations and imaging findings). These patients have collected two different samples of alveolar lavage fluid (BALF) and sputum and have undergone metagenomic next generation sequencing (mNGS) and routine pathogen detection, respectively.
  Interventions: Diagnostic Test: next generation sequencing

INTERVENTIONS:
Diagnostic Test: next generation sequencing — All the enrolled patients had undergone fiberbronchoscopy and sputum had been retained. The collected alveolar lavage fluid and sputum were examined for mNGS and routine etiology, respectively
  Other Names: mNGS

SUMMARY:
Retrospective analysis of clinical data from 50 hospital-admitted patients with suspected pulmonary infection (as judged by clinical manifestations and imaging findings) was performed on study participants who had collected two different samples of alveolar lavage fluid (BALF) and sputum and underwent metagenomic next generation sequencing (mNGS) and routine pathogen detection, respectively. The positive rate of pathogen detection and the consistency of pathogen detection results of the two detection methods were compared to evaluate the clinical manifestation and role of mNGS in pathogen diagnosis.

DETAILED DESCRIPTION:
Pulmonary infection is a common type of respiratory infection that can lead to multiple complications and is considered the most important infectious disease worldwide due to its high morbidity and mortality. Lung infections, caused by one or more pathogens such as bacteria, viruses, fungi and parasites, are not easily distinguishable clinically and are among the top 10 causes of death worldwide. Therefore, early and accurate identification of the cause of infection for patients with pulmonary infection is of great significance for subsequent treatment and improvement of prognosis. At present, the main traditional diagnostic methods for pulmonary infection are microbial culture, antigen and antibody detection and PCR nucleic acid detection technology. Although microbial culture is the gold standard for microbial identification, it takes a long time to detect some viruses and parasites. The sensitivity of antigen and antibody detection is poor. PCR nucleic acid detection method has high sensitivity and specificity, but it can not detect all pathogens causing lung infection. Therefore, it is necessary to develop a fast, convenient and sensitive new detection technology to detect the pathogen of pulmonary infection. next generation sequencing (NGS) has the advantage of no assumptions and no dependence on culture, and can detect all pathogens in clinical samples without bias, and has been widely used in a variety of infectious diseases. This study collected the basic information of patients suspected of pulmonary infection in clinic, and conducted mNGS detection and routine pathogen detection on different samples of alveolar lavage fluid (BALF) and sputum, respectively, to evaluate the consistency of mNGS detection and routine detection and the positive pathogen detection rate, as well as the clinical application value of mNGS detection.

This study retrospectively analyzed 50 patients hospitalized in our hospital from January, 2019 to October, 2019, whose symptoms, signs, imaging and infection indicators met the diagnostic criteria for pulmonary infection, while routine etiological detection of sputum and pulmonary alveolar lavage fluid mNGS were performed.

Clinical data of relevant patients were collected, including gender, age, smoking status, clinical manifestations, length of stay before mNGS detection, antibiotic use before mNGS detection, imaging changes, laboratory examination and other basic information. Results were collected from study participants' alveolar lavage fluid (BALF), sputum for traditional pathogen tests (microbial culture and PCR nucleic acid detection techniques), and mNGS tests. The positive rate of pathogen detection and the consistency of detection results of the two detection methods were compared.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria: Patients meeting diagnostic criteria for pulmonary infection between January 1, 2020 and October 31, 2023. Patients with pulmonary infection were diagnosed with new or worsening focal or diffuse infiltrating lesions on chest CT accompanied by at least one of the following four pneumonic-related clinical manifestations: (1) Recent cough, sputum, or aggravation of existing respiratory symptoms with or without purulent sputum, chest pain, dyspnea, and hemoptysis; ② Heat, T≥38℃; ③ Signs of lung consolidation and/or smell and moist rales; ④ Peripheral blood white blood cell count > 10*109/L or < 4*109/L.

Exclusion criteria: ① The patient did not undergo bronchoscopy; Absence of clinical or laboratory data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose symptoms, signs, imaging, and infection indicators met the diagnostic criteria for pulmonary infection while routine etiological detection of sputum and pulmonary alveolar lavage fluid mNGS were performed.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Etiological detection rates of two detection techniques | From January 1, 2020 to October 31, 2023
  Study participants who had collected two different samples of alveolar lavage fluid (BALF) and sputum and underwent metagenomic next generation sequencing (mNGS) and routine pathogen detection, respectively, compared the positive rates of pathogen detection by the two detection methods

SECONDARY OUTCOMES:
Consistency of detection results of two detection techniques | From January 1, 2020 to October 31, 2023
  Study participants who had collected two different samples of alveolar lavage fluid (BALF) and sputum and underwent metagenomic next generation sequencing (mNGS) and routine pathogen detection, respectively, were compared for the consistency of pathogen detection results between the two assays

CONTACTS AND LOCATIONS:
Overall Officials: Yunfeng Hou, master, Study Director — Department of Intensive Care Medicine, Qiandfo Mountain Hospital, Shandong Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qian YY, Wang HY, Zhou Y, Zhang HC, Zhu YM, Zhou X, Ying Y, Cui P, Wu HL, Zhang WH, Jin JL, Ai JW. Improving Pulmonary Infection Diagnosis with Metagenomic Next Generation Sequencing. Front Cell Infect Microbiol. 2021 Jan 26;10:567615. doi: 10.3389/fcimb.2020.567615. eCollection 2020. PMID 33585263
- [Background] Langelier C, Kalantar KL, Moazed F, Wilson MR, Crawford ED, Deiss T, Belzer A, Bolourchi S, Caldera S, Fung M, Jauregui A, Malcolm K, Lyden A, Khan L, Vessel K, Quan J, Zinter M, Chiu CY, Chow ED, Wilson J, Miller S, Matthay MA, Pollard KS, Christenson S, Calfee CS, DeRisi JL. Integrating host response and unbiased microbe detection for lower respiratory tract infection diagnosis in critically ill adults. Proc Natl Acad Sci U S A. 2018 Dec 26;115(52):E12353-E12362. doi: 10.1073/pnas.1809700115. Epub 2018 Nov 27. PMID 30482864
- [Background] Shi CL, Han P, Tang PJ, Chen MM, Ye ZJ, Wu MY, Shen J, Wu HY, Tan ZQ, Yu X, Rao GH, Zhang JP. Clinical metagenomic sequencing for diagnosis of pulmonary tuberculosis. J Infect. 2020 Oct;81(4):567-574. doi: 10.1016/j.jinf.2020.08.004. Epub 2020 Aug 5. PMID 32768450
- [Background] Yan L, Sun W, Lu Z, Fan L. Metagenomic Next-Generation Sequencing (mNGS) in cerebrospinal fluid for rapid diagnosis of Tuberculosis meningitis in HIV-negative population. Int J Infect Dis. 2020 Jul;96:270-275. doi: 10.1016/j.ijid.2020.04.048. Epub 2020 Apr 24. PMID 32339718
- [Background] Wilson MR, Sample HA, Zorn KC, Arevalo S, Yu G, Neuhaus J, Federman S, Stryke D, Briggs B, Langelier C, Berger A, Douglas V, Josephson SA, Chow FC, Fulton BD, DeRisi JL, Gelfand JM, Naccache SN, Bender J, Dien Bard J, Murkey J, Carlson M, Vespa PM, Vijayan T, Allyn PR, Campeau S, Humphries RM, Klausner JD, Ganzon CD, Memar F, Ocampo NA, Zimmermann LL, Cohen SH, Polage CR, DeBiasi RL, Haller B, Dallas R, Maron G, Hayden R, Messacar K, Dominguez SR, Miller S, Chiu CY. Clinical Metagenomic Sequencing for Diagnosis of Meningitis and Encephalitis. N Engl J Med. 2019 Jun 13;380(24):2327-2340. doi: 10.1056/NEJMoa1803396. PMID 31189036
- [Background] Fida M, Wolf MJ, Hamdi A, Vijayvargiya P, Esquer Garrigos Z, Khalil S, Greenwood-Quaintance KE, Thoendel MJ, Patel R. Detection of Pathogenic Bacteria From Septic Patients Using 16S Ribosomal RNA Gene-Targeted Metagenomic Sequencing. Clin Infect Dis. 2021 Oct 5;73(7):1165-1172. doi: 10.1093/cid/ciab349. PMID 33893492